CLINICAL TRIAL: NCT00984100
Title: Natural Orifice Translumenal Endoscopic Surgery (NOTES) Transvaginal Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baystate Medical Center (Other)
Responsible Party: Principal Investigator, John Romanelli, MD, Baystate Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-086
Record Dates: First submitted 2009-09-23; First posted 2009-09-25 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Cholelithiasis; Biliary Dyskinesia
Keywords: Cholelithiasis; Biliary dyskinesia
MeSH Terms: conditions — Cholelithiasis; Biliary Dyskinesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Notes Transvaginal Cholecystectomy (Experimental): Patients who undergo a NOTES Transvaginal cholescystectomy.
  Interventions: Procedure: NOTES Transvaginal Cholecystectomy

INTERVENTIONS:
Procedure: NOTES Transvaginal Cholecystectomy — An operation to remove the gallbladder, but instead of removing it via an incision in the abdominal wall, will be removed using an endoscope inserted through an opening in the posterior vagina (which then enters the abdominal cavity).

SUMMARY:
Natural Orifice Translumenal Endoscopic Surgery (NOTES) describes a new field of investigational surgery which uses the endoscope as the primary operative tool. The insertion sites for the endoscope include natural orifices such as the mouth, anus, vagina, or urethra. Multidisciplinary teams of surgeons and gastroenterologists collaborate to develop safe and effective surgical techniques via the natural orifice route in order to avoid surgical incisions. Early studies have focused on transvaginal surgery as the access route to the abdomen as it sidesteps troubling questions about infection and closure of the organ. This study is a pilot study to test the feasibility to NOTES transvaginal cholecystectomy using conventional surgical and endoscopic tools.

DETAILED DESCRIPTION:
Introduction: Natural Orifice Translumenal Endoscopic Surgery (NOTES) describes a new field of investigational surgery which uses the endoscope as the primary operative tool. The insertion sites for the endoscope include natural orifices such as the mouth, anus, vagina, or urethra. Multiple animal studies utilizing similar techniques are ongoing at several institutions, including Baystate Medical Center. These multidisciplinary teams consist of surgeons and gastroenterologists who are collaborating to develop safe and effective surgical techniques via the natural orifice route in order to avoid surgical incisions.

The NOTES team at Baystate began animal studies in May, 2006. Multiple procedures, including but not limited to uterine horn resection (simulating appendectomy), cholecystectomy, nephrectomy, splenectomy, distal pancreatectomy, small bowel resection, mediastinal exploration, and sleeve gastrectomy have been completed successfully by the team. This work has led to a separate, IRB-approved protocol to perform NOTES pancreatic pseudocystgastrostomy in human patients. To date, 2 patients have successfully undergone entirely transluminal, endoscopic cystgastrostomy with a third case upcoming. The focus of much of our research (as well as that of many other investigators), is to develop a secure closure method for the stomach. Unfortunately, key scientific questions remain regarding this technique and thus have limited human trials to date. Given this, we have begun to explore other access techniques.

Gynecologists have long considered transvaginal access to the peritoneum as a safe route of entry into the abdomen. Transvaginal hysterectomy and transvaginal tubal ligation have indeed become a regular part of the gynecologic armamentarium. NOTES surgeons have learned from this access approach and have begun to employ it as a safe route into the abdomen. In fact, investigators in New York1,2; San Diego3; Strasbourg, France4; Mallorca, Spain5; Hamburg, Germany6, Milan, Italy7; and Rio de Janeiro8,9 and São Paulo10, Brazil have all announced transvaginal NOTES procedures involving the gallbladder. All of these approaches, to date, have utilized one or more laparoscopic trocars for safety reasons.

Primary Objective: The primary objective of this pilot study is to demonstrate that the Natural Orifice Translumenal Endoscopic Surgery (NOTES) transvaginal cholecystectomy technique is as safe and effective as standard laparoscopic surgical technique for the resection of gallbladder.

Hypothesis: Patients who undergo Natural Orifice Translumenal Endoscopic Surgery for treatment of their gallbladder disease will experience effective treatment with less discomfort and with quicker recovery than standard surgical techniques.

Introduction: The NOTES team (surgeon and gastroenterologist) at Baystate has extensive experience with animal work in developing novel techniques with commercially available products. Despite performing cholecystectomies in porcine models both through a transgastric and transvaginal approach, we have yet to perform a human case. The surgeons on the team have performed well over a thousand laparoscopic cholecystectomies; the gastroenterologist is a recognized advanced therapeutic endoscopist; and the gynecologist is an expert in transvaginal surgery. We believe that our combination of human experience and animal research will lead to safe attempts to perform the procedure described herein.

Methods: There will be a total of 3 patients undergoing this experimental surgical procedure once meeting all entry criteria and subsequent to obtaining informed consent These patients will be recruited from the Baystate ambulatory surgery clinics.. Preoperative laboratory testing, such as blood work (liver function tests, amylase and lipase, a white blood cell count, and a pregnancy test), as well as ultrasound of the liver to document gallbladder disease will be performed as is the standard for patients undergoing surgical removal of the gallbladder. In this procedure, after the induction of general anesthesia and creation of a culdotomy, a sterile endoscope would be inserted into the vagina and then into the abdomen. Following the insertion of the endoscope, a retraction stitch will be passed through the abdominal wall and into the gallbladder to retract the fundus of the gallbladder in a cephalad direction. A 5-mm trocar will be placed in the umbilicus and will serve two functions: one, to allow for a laparoscope in case the view becomes compromised or substandard; and two, to allow a clip applier to be placed in the abdomen for clipping the cystic artery and cystic duct. Dissection of the gallbladder can commence using endoscopic tools and removal of the specimen will be directly through the culdotomy and out through the vagina. Utilizing this technique, as many as three surgical incisions can be avoided.

Postoperatively, the patient will be kept in the hospital overnight. After discharge, follow-up examination will be conducted at 3-5 days (by telephone), 1 week, and 6 weeks following the procedure to determine the success of the procedure. Longer term follow-up will be determined by the patient's overall condition. For at least the first 3 procedures, a laparoscopic camera will be available on the sterile field and at least one laparoscopic trocar will be employed. As with any operation, we would revert to the next least invasive modality should patient safety and/or degree of difficulty dictate that it be so. In this case, should we encounter difficulties during transvaginal cholecystectomy, we would have a low threshold to revert to laparoscopic cholecystectomy or even to open cholecystectomy as needed.

Safety Monitoring: Due to the novelty of the procedure, safety information will be monitored on a continuous basis. Complications that deviate from expected outcomes from standard laparoscopic cholecystectomy would result in, the study being terminated prematurely or temporarily suspended while we assess the events. A member of the general surgery department will be appointed as a safety monitor and will review all the cases and report to the IRB after the first and third case.

Risks and Benefits: The anticipated risks associated with this type of surgery include:

Bleeding, infection, need for open surgery, bile leak, bile duct injury, and bowel injury. Risks specific to the transvaginal NOTES approach include infection of the vagina, dyspareunia. A vaginal incision has no known adverse effects on either fertility or subsequent childbirth, even within a few weeks of the procedure. The anticipated benefits include a decrease in the amount of pain experienced with laparoscopic cholecystectomy, as well as a more cosmetically acceptable result.

Statistics: As this is a purely descriptive study of feasibility of a new technique, there are no specific statistics to be monitored.

Data Storage: The identifiable data collected will be kept in a locked filing cabinet in the primary investigator's office. Only the PI will have access to this file.

It is anticipated that there will be more similar "natural orifice-type" surgeries in the future for a variety of procedures and a multitude of reasons (no incision, less pain, and less time in the hospital). These surgeries will be some of the first transvaginal cholecystectomies performed in the world.

ELIGIBILITY:
Inclusion Criteria:

1. Adult female (18 years old or over) patients who are able to provide informed consent for this surgical procedure
2. Patients scheduled to undergo non-emergent surgical removal of the gallbladder

Exclusion Criteria:

1. Inability to provide informed consent
2. Patients who have a history of prior pelvic surgery (excluding Caesarian sections, tubal ligations, or non-operative pelviscopy)
3. Patients who have acute cholecystitis, gallstone pancreatitis, or who have had a percutaneous cholecystotomy tube placed
4. Patients with a BMI > 40 kg/m2
5. Pregnancy
6. Male gender
7. History of PID

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Morbidity | One year

SECONDARY OUTCOMES:
Mortality | One year
Postoperative pain | One year

CONTACTS AND LOCATIONS:
Overall Officials: John Romanelli, MD, Principal Investigator — Baystate Medical Center
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States